CLINICAL TRIAL: NCT00415961
Title: Multi-Center Clinical Trial: Evaluation of Effectiveness and Safety
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Conor Medsystems (Industry)
Collaborators: Getz Pharma (Industry)
Responsible Party: Shigeru Saito, MD, ShonanKamakura General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-CMS-005
Record Dates: First submitted 2006-12-22; First posted 2006-12-27 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Coronary Disease
Keywords: Percutaneous Coronary Intervention (PCI); Drug-eluting stent (DES)
MeSH Terms: conditions — Coronary Disease

ARMS (1):
- 1 (Experimental): CoStar Paclitaxel drug eluting stent
  Interventions: Device: CoStar Paclitaxel Drug-Eluting Coronary Stent System

INTERVENTIONS:
Device: CoStar Paclitaxel Drug-Eluting Coronary Stent System — CoStar Paclitaxel Drug-Eluting Coronary Stent System

SUMMARY:
This trial aims to demonstrate the non-inferiority of the CI-CMS-005 Coronary Stent System to the study device as well as to the TAXUS™ Express2™ Drug-Eluting Coronary Stent System in in-segment late lumen loss at 9 months after treatment of a single de novo lesion per vessel.

DETAILED DESCRIPTION:
This is a complementary, multi-center, open-label, single-arm trial investigating angiographic and clinical patient outcomes in Japan. Historical data from the 2-arm randomized COSTAR II trial will be used for comparison.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

* Eligible for percutaneous coronary intervention (PCI)
* Documented stable or unstable angina pectoris (Class I, II, III or IV), documented ischemia, or documented silent ischemia
* Documented LVEF ≥25% within the last 6 weeks.
* Eligible for coronary artery bypass graft surgery (CABG)

Exclusion Criteria:

General Exclusion Criteria: -

* Known sensitivity to paclitaxel or polymeric matrices.
* Planned treatment with any other PCI device in the target vessel(s).
* MI within 72 hours prior to the index procedure
* Patient is in cardiogenic shock
* Cerebrovascular Accident (CVA) within the past 6 months
* Acute or chronic renal dysfunction (creatinine >2.0 mg/dl or >150 µmol/L)
* Contraindication to ASA or to ticlopidine
* Thrombocytopenia
* Active GI bleeding within past three months
* Known allergy to cobalt chromium
* Any prior true anaphylactic reaction to contrast agents

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-11; Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
In-segment late lumen loss at 9 months, as measured by QCA. | 9 months

SECONDARY OUTCOMES:
Device, lesion and procedure success; MACE at 30 days and 8 months, Angiographic restenosis at 9 months; Clinically driven Target Lesion Revascularization at 8 months | MACE at 30 days and 8 months, Angiographic restenosis at 9 months; Clinically driven Target Lesion Revascularization at 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Saito, MD, Principal Investigator — ShonanKamakura General Hospital
Locations (1):
- Shonan Kamakura General Hospital, Kamakura, Japan